CLINICAL TRIAL: NCT02165462
Title: Assessment of Bilateral Deficit Phenomenon During Dynamic Plantar Flexion Task in Patients With Haemophilic Arthropathy
Brief Title: Bilateral Deficit Phenomenon in Patients With Haemophilic Arthropathy
Acronym: PROPRIO-HE
Status: Completed | Type: Observational
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Rubén Cuesta-Barriuso, PhD, PhD, Universidad Católica San Antonio de Murcia
Other Study IDs: PROPRIO-HE
Record Dates: First submitted 2014-06-01; First posted 2014-06-17 (Estimated); Results first posted 2015-12-15 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2015-09

CONDITIONS: Hemophilia
Keywords: Haemophilia; Arthropathy; Bilateral deficit phenomenon; Proprioception
MeSH Terms: conditions — Hemophilia A; Joint Diseases | interventions — hydroxyethyl methacrylate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with haemophilia: Assessment of bilateral deficit phenomenon during dynamic plantar flexion task
  Interventions: Other: Patients with haemophilia

INTERVENTIONS:
Other: Patients with haemophilia — Assessment of bilateral deficit phenomenon during dynamic plantar flexion task with a force platform (Kistler 9286 BA model, Kistler Instruments, Amherst, NY, USA)

SUMMARY:
Trial to assess the bilateral deficit phenomenon during dynamic plantar flexion task in patients with haemophilic arthropathy Describe the differences in terms of the physical variables (muscular strength, range of motion and proprioception) in patients with hemophilia who have conducted a home treatment with a digital tool.

Bookmark the relationship between clinical history of joint bleeds and clinical manifestations in standing and walking.

DETAILED DESCRIPTION:
* Assess the bilateral deficit phenomenon during dynamic plantar flexion task in patients with haemophilic arthropathy.
* Indicate the independent variables that influence the development of strength and contractile activity, with or without previous joint bleeds in haemophilia patients with minors.
* Observe the descriptive variables people influence the standing, the incorporation from sitting and jumping.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with hemophilia A and B.
* With or without joint involvement clinically diagnosed, and with or without a previous history of hemarthrosis joint load legs.
* In prophylactic regimen with FVIII / FIX concentrates .
* Residents in the Autonomous Community of the Region of Murcia.

Exclusion Criteria:

* Patients without walking ability.
* Patients diagnosed with other congenital coagulopathy (von Willebrand disease, etc..).
* Patients with neurological or cognitive impairments that prevent understanding the questionnaires and physical tests.
* Patients whose parents or guardians have not signed the informed consent document.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with haemophilia
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2015-09; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: JUAN JOSE RODRIGUEZ, MsC, Study Chair — Universidad Católica San Antonio; RUBEN CUESTA-BARRIUSO, PhD, Principal Investigator — Universidad Católica San Antonio
Locations (1):
- Universidad Católica San Antonio, Murcia, Murcia, Murcia, Spain

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with haemophilia
Period: Overall Study
Arm/Group | Patients With Haemophilia
Started | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients With Haemophilia
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.47 (7.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 17
Region of Enrollment [Number; unit: participants]
  Spain | 17

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Bilateral Index of Maximal Peak Force
Description: Assessment of bilateral index of maximal peak force with a force platform (Kistler 9286 BA model, Kistler Instruments, Amherst, NY, USA).
Time Frame: Screening visit
Population: Bilateral rates was calculated during the preparation phase and during the acceleration phase to express relative difference in strength between bilateral and unilateral conditions. Based on information in the Howard and Enoka (1991), the calculation detail for the Bilateral Index is "[100x (bilateral) / (right unilateral + left unilateral)] - 100"
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Patients With Haemophilia
Number analyzed (Participants) | 17
percentage | -40.86 (4.24)

2. Primary Outcome: Assessment of Bilateral Index of Rate of Development During the Preparation Phase
Description: Assessment of Bilateral index of rate of development during the preparation phase with a force platform (Kistler 9286 BA model, Kistler Instruments, Amherst, NY, USA)
Time Frame: Screening visit
Population: Bilateral rates was calculated during the preparation phase to express relative difference in strength between bilateral and unilateral conditions (calculated in percentages). Based on information in the Howard and Enoka (1991), the calculation detail for the Bilateral Index is "[100x (bilateral) / (right unilateral + left unilateral)] - 100"
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Patients With Haemophilia
Number analyzed (Participants) | 17
percentage | 31.34 (56.42)

3. Primary Outcome: Assessment of Bilateral Index of Rate of Development During the Acceleration Phase
Description: Assessment of bilateral index of rate of development during the acceleration phase with a force platform (Kistler 9286 BA model, Kistler Instruments, Amherst, NY, USA)
Time Frame: Screening visit
Population: Bilateral rates was calculated during the acceleration phase to express relative difference in strength between bilateral and unilateral conditions (calculated in percentages). Based on information in the Howard and Enoka (1991), the calculation detail for the Bilateral Index is "[100x (bilateral) / (right unilateral + left unilateral)] - 100"
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Patients With Haemophilia
Number analyzed (Participants) | 17
percentage | 20.05 (38.20)

4. Primary Outcome: Assessment of Maximal Peak Force
Description: Assessment of maximal peak force with a force platform (Kistler 9286 BA model, Kistler Instruments, Amherst, NY, USA)
Time Frame: Screening visit
Population: The maximum peak force (MPF) is defined as the maximum achieved in the force-time curve during the dynamic test plantar flexion for both bilateral conditions as right and left unilateral, normalized to body weight of the participants (N / kg value)
Measure: Mean (Standard Deviation); unit: N/kg
Arm/Group | Patients With Haemophilia
Number analyzed (Participants) | 17
N/kg | 15.67 (1.36)

5. Primary Outcome: Assessment of Rate of Development During the Preparation Phase
Description: Assessment of rate of development during the preparation phase with a force platform (Kistler 9286 BA model, Kistler Instruments, Amherst, NY, USA)
Time Frame: Screening visit
Measure: Mean (Standard Deviation); unit: N/s
Arm/Group | Patients With Haemophilia
Number analyzed (Participants) | 17
N/s | 6190.86 (2818.36)

6. Primary Outcome: Change of Joint Condition Based on Clinical Assessment
Description: Spanish version of the Haemophilia Joint Health Score 2.1 (HJHS). Additive scale that assesses from 0 to 24 points joint status of patients with haemophilia (0: no joint damage; 24: maximum joint damage).
  The variables studied in this scale are: Swelling (range 0-3); Duration of swelling (range 0-1); Muscle atrophy (range 0-2); Crepitant in motion (range 0-2); Loss of Flexion (range 0-3); Loss of extension (range 0-3); Joint pain (range 0-2): Strength (range 0-4); Gait (range 0-4)
Time Frame: Screening visit
Measure: Mean (Standard Deviation); unit: Units on a scale (range 0-24)
Arm/Group | Patients With Haemophilia
Number analyzed (Participants) | 17
Units on a scale (range 0-24)
  Right knee | 4.88 (4.076)
  Left knee | 3.00 (2.398)
  Right ankle | 5.82 (3.575)
  Left ankle | 6.35 (4.527)

7. Primary Outcome: Assessment of Rate of Development During the Acceleration Phase
Description: Assessment of rate of development during the acceleration phase with a force platform (Kistler 9286 BA model, Kistler Instruments, Amherst, NY, USA)
Time Frame: Screening visit
Measure: Mean (Standard Deviation); unit: N/s
Arm/Group | Patients With Haemophilia
Number analyzed (Participants) | 17
N/s | 8945.25 (2807.85)

8. Primary Outcome: Assessment of Maximal Velocity of Movement
Description: Assessment of maximal velocity of movement with a force platform (Kistler 9286 BA model, Kistler Instruments, Amherst, NY, USA)
Time Frame: Screening visit
Population: The maximum speed (Vmax) was calculated as the maximum value of the first integral of the force-time curve for bilateral contractions, left-sided and right-sided
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Patients With Haemophilia
Number analyzed (Participants) | 17
m/s | 0.48 (0.11)

9. Secondary Outcome: Weight of the Patients With Haemophilia
Description: The weight were collected using a TANITA equipment (TBF-300WA model, Tanita Corporation of America, Inc., Illinois, USA)
Time Frame: Screening visit
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Patients With Haemophilia
Number analyzed (Participants) | 17
Kg | 73.48 (15.43)

10. Secondary Outcome: Diagnosis, Severity of Hemophilia, Treatment (Prophylactic or on Demand)
Description: Patients fill out a registration key clinical data (type, severity of hemophilia, hemarthrosis in the previous month and current drug therapy).
Time Frame: Screening visit
Measure: Number; unit: participants
Arm/Group | Patients With Haemophilia
Number analyzed (Participants) | 17
participants
  Haemophilia A | 15
  Haemophilia B | 2
  Severe haemophilia | 7
  Moderate haemophilia | 5
  Mild haemophilia | 5
  Prophylaxis treatment | 8
  On demand treatment | 9

11. Secondary Outcome: Joint Bleeding Before the Assessment
Time Frame: Screening visit
Measure: Number; unit: participants
Arm/Group | Patients With Haemophilia
Number analyzed (Participants) | 17
participants | 7

12. Secondary Outcome: Height of the Patients With Haemophilia
Description: The height of patients was calculated using a TANITA equipment (TBF-300WA model, Tanita Corporation of America, Inc., Illinois, USA).
Time Frame: Screening visit
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Patients With Haemophilia
Number analyzed (Participants) | 17
cm | 176.53 (6.82)

13. Secondary Outcome: Body Mass Index of Patients With Haemophilia
Description: The body mass index of patients was calculated using a TANITA equipment (TBF-300WA model, Tanita Corporation of America, Inc., Illinois, USA).
Time Frame: Screening visit
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | Patients With Haemophilia
Number analyzed (Participants) | 17
kg/m2 | 23.36 (4.48)

14. Secondary Outcome: Age of Patients With Haemophilia
Time Frame: Screening visit
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Patients With Haemophilia
Number analyzed (Participants) | 17
years | 32.47 (7.82)

ADVERSE EVENTS:
Description: Adverse Events were not collected/assessed
Arm/Group | Patients With Haemophilia
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No